CLINICAL TRIAL: NCT07265362
Title: Compassion Focussed Therapy Informed Psychoeducation and Loving Kindness Meditation for Children and Young People With Epilepsy
Brief Title: Compassion Focussed Therapy Informed Psychoeducation and Loving Kindness Meditation for Young People With Epilepsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 353407
Record Dates: First submitted 2025-07-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Mental Health; Children
Keywords: Epilepsy; Compassion Focussed Therapy; Children; Young People; Teenagers; Mental health; Shame; Self-compassion; Loving Kindness Meditation
MeSH Terms: conditions — Epilepsy; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion Focussed Therapy and Loving Kindness Meditation Intervention (Experimental): Single arm study
  Interventions: Other: Compassion Focussed Therapy/Loving Kindness Meditation

INTERVENTIONS:
Other: Compassion Focussed Therapy/Loving Kindness Meditation — After a baseline of 3-5 weeks (randomly allocated) is completed, the participant will engage in three sessions of Compassion Focussed Therapy informed psycho-education and introduction to Loving Kindness Meditation (LKM). Following the third session, the participants will have four weeks to practice LKM, receiving weekly email reminders with guided self-help instructions and reminders to complete outcome measures. A final follow-up session will occur after the four weeks, to consolidate knowledge and skills with the participant, plus gather feedback on the intervention.

SUMMARY:
It has frequently been shown that people with long term physical health conditions, like epilepsy, are more likely to have mental health conditions. Studies have shown people with epilepsy report high levels of shame, stress, social isolation and anxiety. Mental health interventions for people with epilepsy, particularly children, has been identified as an area for further research by the NHS.

Compassion based interventions have been effective with people with long term physical health conditions. These interventions aim to develop an individual's compassion towards the self and others in response to self-criticism or shame. This study aims to explore whether Compassion Focussed Therapy informed psychoeducation and Loving Kindness Meditation is a feasible and effective intervention for children with epilepsy.

Children and young people aged 12-17 years old who have a diagnosis of epilepsy and mild/moderate distress related to their health condition are eligible. Local clinicians in epilepsy services will be asked to identify potential participants. Up to six children/young people will be included in the study. Participants will complete outcomes measures (about their quality of life, mood and self-compassion) weekly before the intervention, for up to five weeks, and then weekly until the end of the intervention. The intervention will be three sessions with the lead researcher, conducted online via Microsoft teams. Participants will then have four weeks to practice Loving Kindness Meditation. They will then have a follow up session about how they found the intervention, what was helpful and what they would change. The results from the study will indicate whether Compassion Focussed Therapy and Loving Kindness Meditation is a beneficial therapeutic intervention for children with epilepsy and if further research in the area is warranted.

DETAILED DESCRIPTION:
Of the 533,000 people in England and Wales with epilepsy, 112,000 are children and young people (National Institute for Health and Care Excellence, 2022). The reported rates of diagnosed mental health conditions in children with epilepsy (CWE) vary significantly across studies, from 30% to 70% (NHS England, 2024; Young Epilepsy, 2021), but it is consistently found that CWE are more likely to have mental health difficulties than their peers, including depression, anxiety, low self-esteem and stress (Ekinci et al., 2009; Chew et al., 2019; Batchelor & Taylor, 2021; Stefanidou et al., 2020). Negative daily life events, such as experiencing stigma, social exclusion, and limited understanding from professionals and peers, are just some of the stressors reported by CWE (Benson et al., 2016; Stefanidou et al., 2020; Young Epilepsy, 2021; Moffat et al., 2009). A scoping review found parents and caregivers also have concerns about the mental health of their CWE, including worrying they will have negative self-image and reduced social activity (Carter et al., 2022). Epilepsy has been recognised as one of the key areas for change for children and young people by NHS England's Core20PLUS5 approach (NHS England, 2022). Adolescence has been identified as a significant period for those with epilepsy, with stressors like transition to adult services (Stefanidou et al., 2020) increasing the prevalence of mental health issues. Studies suggest that treatment for epilepsy needs to take a holistic approach (Healy et al., 2020) and include mental health as an important factor in treatment and screening at epilepsy diagnosis (Wagner et al., 2016). People with epilepsy have been shown to have higher rates of shame and self-disgust than the general population (Räty et al., 2009; Mayor et al., 2022a; Mayor et al., 2022b). Shame has been linked with the unfortunate, ongoing stigma around epilepsy (Morrell, 2002; Şengül & Kurudirek, 2022). The double stigma phenomenon is when a person has dual conditions that are stigmatised in society (e.g. epilepsy and mental health issues; Mula & Kaufman, 2020). The phenomenon as applied to epilepsy suggests that perceived stigma from others also leads to feelings of shame for people with epilepsy, in turn increasing the prevalence of mental health issues (Bandstra et al., 2008; Henning et al., 2021). Baker et al.'s (2018) systematic review found increased stigma led to reduce psychological wellbeing. CWE as young as nine years old have been found to be affected by stigma (Austin et al., 2014). Stigma and shame are IRAS Form Reference: 25/EM/0153 IRAS Version 6.4.3 Date: 03/07/2025 353407/1734733/37/270 9 closely linked, with shame particularly associated with increased mental health issues, such as depressive symptoms (Kim et al., 2011). The evidence base for psychological interventions for CWE has been growing in recent years (Mercier & Dorris, 2024), but few interventions appear to target the unique experience of shame within epilepsy. Some mental health interventions have been identified for people with epilepsy. A Cochrane review (Michaelis et al., 2020) found moderate evidence for skills-based interventions for people with epilepsy, such as Cognitive Behavioural Therapy (CBT) and mindfulness-based interventions. However, it can often be difficult for people with epilepsy to access mental health support, for reasons such as availability and accessibility (Mahendran et al., 2017; Shaw et al., 2019). It has been recognised that the lack of mental health resources for this population is an area needing further research, particularly for CWE (NICE, 2022). One barrier to treatment in the UK is current service provision, which varies across the NHS. Children and young people with long-term health conditions can often be excluded from accessing Child and Adolescent Mental Health Services (CAMHS; Children's Commissioner for England, 2016) and improvements are needed for referral pathways to tertiary paediatric epilepsy services (NHS England, 2024). Recommendations for researching online interventions for people with epilepsy have already been made (NICE, 2022), the benefits of which include cost-effectiveness and accessibility, hence the increase in digital interventions being offered in healthcare. Evidence for online psychological intervention is growing, with meta-analyses showing effectiveness (Spijkerman et al., 2016; Fu et al., 2020). The use of online psychological intervention has also been positively evidenced for people with long-term health conditions, for example, by reducing barriers like the inability to travel due to health (Beatty & Lambert, 2013; White et al., 2020; Lee et al., 2024). Lecce et al.'s (2023) systematic review concluded that digital mental health interventions for people with epilepsy specifically were effective and could improve access to psychological interventions for underserved populations. Digital mental health interventions for young people have also been reviewed and found to be effective (Zhou et al., 2021), although Lehtimaki et al. (2020) suggest more evidence is needed to show consistent effectiveness. Digital mental health interventions for young people with long term health conditions have been developed and tested with promising results of acceptability, feasibility and positive engagement, (Brigden et al., 2020; Palermo et al., 2020; Finlay-Jones et al., 2023). However, other evidence has found that despite feasibility (Ferrario, 2021), the evidence base is heterogenous, and reviews have frequently struggled to ascertain good quality evidence to include (Bennett et al., 2019; Fisher et al., 2019). There have also been identified difficulties in engagement, leading to participant attrition (Voerman et al., 2015). Provision of therapist engagement can increase participation, such as weekly phone calls or emails (Bennett et al., 2019). Self-guided interventions are generally seen to have potential for effectiveness and have been recommended to policy makers (Camp-Spivey et al., 2021; Azevedo et al., 2021), as well as receiving positive feedback on patient satisfaction measures (Bennett et al., 2018; Fisher et al., 2019). Compassion Focussed Therapy (CFT) was introduced by Paul Gilbert (2009). CFT defines compassion as "sensitivity to suffering distress in self and others, with a commitment to try to alleviate and prevent it" (Gilbert et al., 2017). As the focus of CFT is upon shame and self-criticism (Gilbert, 2009), this therapeutic modality aligns with the impacts of epilepsy outlined above. Specific aspects of CFT, such as self-compassion, have been linked with reduced psychological distress and improved wellbeing for people with chronic physical health conditions in cross-sectional studies, meta-analyses and systematic reviews (Clegg et al., 2019; Phillips & Hine, 2021; Kılıç et al., 2021). Baker et al. (2019) found self-compassion to be of possible importance for reducing psychological distress in people with epilepsy specifically. CFT has been effectively used with children previously (Bratt et al., 2020; Carona et al., 2017). Self-compassion based approaches have been found to be effective for CYP with long-term physical health conditions, like diabetes and chronic pain conditions (Jackson, 2018; Prentice et al., 2021). One type of compassionate imagery is Loving Kindness Meditation (LKM; Gilbert, 2010). LKM is a mindfulness practice that has been shown to develop self-compassion by developing unconditional kindness to the self and others (Hofmann et al., 2011). Reilly and Stuyvenberg's (2022) meta-analysis found a moderate overall effect for LKM with adults. A meta-analysis reviewing the effect of LKM for children and adolescents found improvements in wellbeing and concluded that the findings were encouraging, but criticised the quality of the evidence (Perkins et al., 2022). There is also emerging evidence of the impact of LKM on neurobiology and brain structures in long-term practice (Bashir er al., 2025; Wong et al., 2022). As evidence shows that self-compassion based interventions can reduce feelings of shame (Woods & Proeve, 2014; Callow et al., 2021), it therefore appears feasible to test the effects of LKM with a population who have high levels of shame. This project overall aims to add to the limited evidence base that currently exists for mental health interventions for CWE, despite many findings showing that people with epilepsy have a higher likelihood of having mental health issues. There is evidence for CBT and online psychological intervention being beneficial to CWE, but widening the options for mental health intervention with CWE and furthering the evidence base is an important and recognised need in this area. As stated above, the unique experience of perceived stigma and shame in CWE could be well aligned with self-compassion based interventions that address these feelings specifically. A project providing CFT informed psycho-education and guided self-help on LKM for CWE would therefore be utilising a therapy aimed at addressing shame in a population that has high levels of and a unique experience of shame and stigma. Introducing LKM which aims to improve self-compassion, which in turn can alleviate feelings of shame, has the potential to be a beneficial intervention for CWE.

The proposed study will be an effectiveness study using a Single Case Experimental Design (SCED) series. Through a SCED, individual behavioural data can be collected throughout an intervention (Lane & Gast, 2013). A minimum of three participants (as recommended by methodology guidelines; Krasny-Pacini & Evans, 2018) will be recruited from local secondary and tertiary epilepsy NHS services. A maximum sample size of six has been determined due to resource availability for the research and to account for possible attrition. Local clinicians will be provided with the eligibility criteria and participant information sheet to identify potential participants for the study. If potential participants and caregivers consent to the local clinician sharing information, their details will be sent to the researcher. Contact will be made to ascertain consent from parents/caregivers for children under 16 years of age, and assent will be gained from the child. Informed consent will be obtained from the child, for those over 16 years old. Following an initial screening meeting to ensure eligibility by the researcher and complete baseline measures, participants will be randomly allocated to a baseline of three, four or five weeks, completing weekly outcome measures. Participants will be randomised to baselines of various lengths to have a minimum number of data points for a SCED. A multiple baselines design has been chosen as it is not possible to return to baseline following the intervention (Krasny-Pacini & Evans, 2018). Participants will be allocated a baseline of three, four or five weeks. Microsoft Excel will be used to randomise participants to a baseline length. Once randomised, baseline measures will be sent for participants to complete. The measures section states how frequently each measure will be completed. After the baseline is completed, the participant will engage in three sessions of Compassion Focussed Therapy informed psycho-education and introduction to Loving Kindness Meditation (LKM). Following the third session, the participants will have four weeks to practice LKM, receiving weekly email reminders with guided self-help instructions and reminders to complete outcome measures. A final follow-up session will occur after the four weeks, to consolidate knowledge and skills with the participant, plus gather feedback on the intervention. The follow-up session will be completed via Microsoft Teams and be recorded (with participant assent or consent and parent/caregiver consent). Once all participants have completed the follow up session, analysis will be completed.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* Have a diagnosis of epilepsy. This is to be confirmed by the recruiting professional who will confirm via the participant's medical records.
* Currently showing or reporting mild-moderate psychological distress: including anxiety, low mood or stress, in relation to their health condition, as identified by local clinicians recruiting to study.
* Have access to a computer/internet enabled electronic device e.g. a tablet or mobile phone.
* English speaker to a standard sufficient to participate in verbal communication without an interpreter.

Exclusion Criteria:

* Presence of an Intellectual Disability. As this is a time limited intervention with a set protocol, there will not be opportunity to make adaptations to the intervention. Consistency across the participants is important to show any effect of the intervention.
* Currently receiving any other mental health treatment in order to reduce extraneous variables from other mental health treatment.
* Current report of self-harming behaviours as the research cannot monitor or manage risk.
* Severe psychological distress e.g. depression, psychosis or an eating disorder, as this is likely to require specialist psychological support.
* Seizures are due to Non-Epileptic Attack Disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Idiographic shame and self-compassion measures | Weekly from baseline to end of intervnetion (13 to 15 weeks depending on randomly allocated baseline length)
  Idiographic shame and self-compassion weekly measures. Idiographic measures can be designed to ensure the relevant construct is measured by individual participants (Haynes et al., 2009). In this study, utilising idiographic measures will ensure we measure the constructs of shame and self-compassion more effectively than broader psychometric measures. Possible example shame question: "I have been bothered by other people's reactions to my seizures." Possible example self-compassion question: "I have been kind to myself when something has gone wrong."

SECONDARY OUTCOMES:
Glasgow Epilepsy Outcome Scale for Young Persons (GEOS-YP) | At initial baseline, first week pre-intervention and in the final week after intervention has been complete - week 13, 14 or 15 depending on length of baseline.
  The GEOS-YP was developed by McEwan et al. (2004) in Glasgow, UK. It is a measure of the impact of epilepsy on CYP's quality of life. Adolescents (aged 10 to 18) with a diagnosis of epilepsy co-produced the scale through focus groups and pilot studies, and found good face and content validity. Townshend et al. (2008) found good internal consistency (α = 0.91) and test-retest reliability (p = 0.75). Higher scores indicate better quality of life reported by the CYP. The GEOS-YP will be completed at baseline, pre intervention and at follow up.
PedsQL - parent/caregiver proxy report | At initial baseline, first week pre-intervention and in the final week after intervention has been complete - week 13, 14 or 15 depending on length of baseline.
  The PedsQL was developed in the US as a measure of health related quality of life. The PedsQL has child and proxy versions that can be completed by parents/caregivers. The PedsQL is divided into age groups - the measures for 8-12 and 13-18 years will both be used in the proposed study. Upton et al. (2005) validated the UK-English version of the PedsQL, both self and proxy measures. The sample for proxy measures was 970 parents of children both with and without chronic health conditions. Varni et al. (2007) showed internal reliability scores of the scale to exceed 0.70 for proxy subscales, as well as demonstrating construct validity with the known groups approach. Upton et al. (2005) concluded the scale performed as well in the UK as the US. High scores indicate better health-related quality of life.
Self-Compassion Scale for Youth | At initial baseline, first week pre-intervention and in the final week after intervention has been complete - week 13, 14 or 15 depending on length of baseline.
  The SCS-Y was developed by Neff et al. (2021). It contains six subscales (Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness and Over-identification) and a total self-compassion score. The SCS-Y was based on an adult version of the scale and first validated for youth in the US. Cheung et al. (2023) validated the SCS-Y with a UK sample of 1104 participants aged 12-18 years old. Good internal consistency (α = 0.88) and concurrent validity (r = 0.84, p < 0.01) were found. High scores indicate greater self-compassion.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Moghaddam, DClinPsy, Principal Investigator — University of Lincoln
Locations (1):
- University of Lincoln, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No